CLINICAL TRIAL: NCT06835764
Title: Enhancing Self-Efficacy and Lowering Anxiety Through a Telenovela Intervention for Caregivers of African-American and Hispanic Hospice Patients
Brief Title: A Telenovela Intervention for Caregivers of African-American and Hispanic Hospice Patients
Acronym: NOVELA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Maryland Cigarette Restitution Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00457633; CRF25 (Other: Maryland Cigarette Restitution Fund Research Grant to JHMI (FY25))
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Hospice; Caregivers
Keywords: videos; hospice family caregivers; education; telenovelas; self-efficacy; anxiety; feasibility
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research staff analyzing data will be unaware of study arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOVELA (Experimental): Hospice family caregivers will work with the interventionist to use a web-enabled device (computer, smartphone or tablet) to access and view the video (3-6 mins) over the course of 4 hospice telehealth visits, twice per week.
  Interventions: Behavioral: NOVELA
- Usual hospice care (No Intervention): HFCGs will receive usual hospice care.

INTERVENTIONS:
Behavioral: NOVELA — The family caregivers that consent to participate will work with the interventionist to use a web-enabled device (computer, smartphone or tablet) to access and view the telenovela video (one of four episodes, each 3-6 mins) twice per week over the course of 4 hospice telehealth visits (one episode per visit). All four visits will use telehealth via video-conferencing. The number of visits is based on the number of videos which content is prioritized based on previous work. The interventionist will introduce the purpose and topic of the video, facilitate video viewing and then elicit clarifying questions and reinforce main message.
  Arms: NOVELA

SUMMARY:
This randomized clinical trial (RCT) intends to look at the preliminary efficacy of NOVELA (intervention group) in changing anxiety and self-efficacy compared to usual hospice care (control group). In the NOVELA intervention, hospice care will be enhanced with the telenovela videos for hospice family caregivers (HFCG) education during twice weekly hospice telehealth visits to prepare caregivers for proper use of hospice support and healthcare services.

DETAILED DESCRIPTION:
Telenovela is a television drama or soap opera that can be used to lead viewers to contemplate and discuss critical issues through video storytelling. Prior work showed informational telenovelas had a positive effect on Latino family caregivers' attitudes toward end-of-life (EOL) care services. The role of videos in hospice and palliative care shows significant promise, underscoring the videos as a mode of education for family caregivers that could potentially enhance caregiver's self-efficacy, decrease caregiver's anxiety, and reduce burnout. Despite the value of video education, many programs have failed to provide engaging material.

Based on input from HFCG, the investigators have produced a bilingual (Spanish and English version) four chapter telenovela video series (To Care/ El privilegio de cuidar) as part of NCI funded diversity supplement study. Founded upon extensive preliminary work, To Care portrays the journey of one hospice family as the family struggle with the hospice decision, pain management, decision-making, and finally the dying process. Averaging only 4:65 minutes, each chapter addresses one of these problems, validating family experiences and identifying potential solutions.

In a follow-up study, the investigators developed an interventionist-led conversation guide as a companion for the telenovela. The intervention, which includes the video series and the conversation guide, is named NOVELA (short for telenovela). The investigators preliminary single-arm trial found NOVELA feasible and acceptable in the hospice setting, with promising improvements in caregiver anxiety symptoms. Thus, storytelling and culturally tailored videos can be powerful tools to educate family caregivers of hospice patients. The overall expectation is that NOVELA will improve self-efficacy thus lowering anxiety in hospice family caregivers.

This proposal has the following aims:

* Specific Aim 1: Investigate the preliminary efficacy of delivering NOVELA to African American (AA) and Hispanic HFCGs of cancer patients.
* Specific Aim 2: Evaluate the benefits of NOVELA as perceived by hospice staff.

ELIGIBILITY:
Inclusion Criteria:

* Identified family caregiver of patients enrolled in hospice
* Caregivers must be over the age of 18
* Without cognitive impairment
* With access to wireless device and internet.

Exclusion Criteria:

* HFCG of patients that are actively dying
* Caregivers younger than 18 years
* With cognitive impairment
* Without internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in HFCG Anxiety before and after NOVELA as assessed by the Generalized Anxiety Disorder 7-item scale | Baseline and 2 weeks
  Generalized Anxiety Disorder 7-item (GAD-7) scale. Family caregiver indicate the frequency participants have been bothered by generalized anxiety. 7-items, scale 0-3, score range 0-21; higher scores reflect higher anxiety.
Change in HFCG Self-efficacy before and after NOVELA as assessed by the Caregiver Self-Efficacy Scale | Baseline and 2 weeks
  Caregiver Self-Efficacy Scale (CaSES) - 21-items, scale 1-4, score range 21-84; higher scores reflect higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: DULCE CRUZ-OLIVER, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Univeristy, Baltimore, Maryland, United States

REFERENCES:
- [Background] Crist JD, Pasvogel A, Hepworth JT, Koerner KM. The impact of a telenovela intervention on use of home health care services and Mexican American older adult and caregiver outcomes. Res Gerontol Nurs. 2015 Mar-Apr;8(2):62-76. doi: 10.3928/19404921-20150105-02. Epub 2015 Jan 16. PMID 25594360
- [Background] Cruz-Oliver DM, Malmstrom TK, Fernandez N, Parikh M, Garcia J, Sanchez-Reilly S. Education Intervention "Caregivers Like Me" for Latino Family Caregivers Improved Attitudes Toward Professional Assistance at End-of-life Care. Am J Hosp Palliat Care. 2016 Jul;33(6):527-36. doi: 10.1177/1049909115584315. Epub 2015 May 27. PMID 26019262
- [Background] Washington KT, Oliver DP, Benson JJ, Rolbiecki AJ, Jorgensen LA, Cruz-Oliver DM, Demiris G. Factors influencing engagement in an online support group for family caregivers of individuals with advanced cancer. J Psychosoc Oncol. 2020 May-Jun;38(3):235-250. doi: 10.1080/07347332.2019.1680592. Epub 2019 Nov 6. PMID 31690247
- [Background] Cruz-Oliver DM, Abshire M, Budhathoki C, Oliver DP, Volandes A, Smith TJ. Reflections of Hospice Staff Members About Educating Hospice Family Caregivers Through Telenovela. Am J Hosp Palliat Care. 2021 Feb;38(2):161-168. doi: 10.1177/1049909120936169. Epub 2020 Jul 8. PMID 32638608